CLINICAL TRIAL: NCT00846118
Title: Differential Intervention Trial by Standard Therapy Versus Pitavastatin in Patients With Chronic Hemodialysis.
Brief Title: Differential Intervention Trial by Standard Therapy Versus Pitavastatin in Patients With Chronic Hemodialysis (DIALYSIS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Chieko Hamada (Other)
Responsible Party: Sponsor-Investigator, Chieko Hamada, Division of Nehprology, Juntendo University
Organization: Juntendo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208-032
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Disease
Keywords: Pitavastatin; Hemodialysis; Mortality; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitavastatin (Active Comparator): Pitavastatin in addition to optimal standard care
  Interventions: Drug: Pitavastatin
- optimal standard care (No Intervention)

INTERVENTIONS:
Drug: Pitavastatin — 1-4mg/day
  Other Names: LIVALO
  Arms: Pitavastatin

SUMMARY:
The purpose of this study is to verify whether pitavastatin prevents from cardiovascular events and improves the mortality in chronic hemodialysis patients with hypercholesteremia.

DETAILED DESCRIPTION:
It was already proved by the clinical trials that statins prevent from death and cardiovascular events. However, the efficacy of statins in patients with chronic hemodialysis has not been proved yet.

ELIGIBILITY:
Inclusion Criteria:

* patients under hemodialysis
* patients with hypercholesterolemia as defined by any of following parameters:

  * LDL-C ≧ 100 mg / dL
  * TC ≧ 180 mg / dL
  * patients required cholesterol-lowering treatment by investigators.
* patients aged 20-75 years
* patients with written consent by their own volition after being provided sufficient explanation for the participation into this clinical trial

Exclusion Criteria:

* patients taking statins or fibrates
* patients enrolled to the other trials using contraindication drugs of pitavastatin
* patients who had acute myocardial infarction within six months before the day of the agreement acquisition
* patients scheduled PCI and CABG within six months after the day of the agreement acquisition
* Patients who had diagnosis or doubt of malignant tumor
* patients corresponded to "Contraindications" of pitavastatin
* Familial hypercholesterolemia patients
* patients judged ineligible by investigators

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2011-01-31 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
all cause mortality | whole observational period
Myocardial infarction of the new onset | whole observational period

SECONDARY OUTCOMES:
Cardiac death | whole observational period
Myocardial infarction of the new onset | whole observational period

OTHER OUTCOMES:
interventions for ischemic heart disease | whole observational period
Serious arrhythmia | whole observational period
Hospitalization for the heart failure | whole observational period
Hospitalization for the unstable angina | whole observational period
cerebral stroke | whole observational period
Bone fracture | whole observational period

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Tomino, MD,PhD, Principal Investigator — Professor of Medicine, Department of Nephrology, Juntendo University Graduate School of Medicine
Locations (1):
- Division of Nephrology, Department of Internal Medicine, Juntendo Hospital, Tokyo, Japan